CLINICAL TRIAL: NCT00059657
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of CirculaseTM in Conjunction With Peripheral Revascularization for the Treatment of Critical Leg Ischemia
Brief Title: Efficacy/Safety of Ecraprost in Lipid Emulsion for Treatment of Critical Leg Ischemia Due to Peripheral Arterial Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WFI 01-02
Record Dates: First submitted 2003-04-29; First posted 2003-05-02 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Peripheral Vascular Disease
Keywords: Ecraprost in lipid emulsion; CLI; peripheral, vascular; amputation; Angioplasty; by-pass; Critical Limb Ischemia due to peripheral arterial disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Ecraprost

INTERVENTIONS:
Drug: Ecraprost in lipid emulsion

SUMMARY:
Ecraprost in lipid emulsion is being developed for the treatment of Critical leg ischemia (CLI), which is the most severe form of peripheral arterial disease (PAD); This trial is designed to assess the efficacy and safety of the drug in the treatment of CLI.

ELIGIBILITY:
Inclusion Criteria:

* Critical leg ischemia (CLI) defined as distal extremity pain at rest, or peripheral ischemic ulcer(s), with severe hemodynamic impairment as diagnosed by ankle systolic pressure, toe systolic pressure or TcPO2
* Subjects will already be scheduled to receive a revascularization procedure (e.g., by-pass graft, endovascular procedure, etc.) involving a distal target artery below the knee joint (e.g., below the knee joint popliteal, anterior/posterior tibial, peroneal, plantar, pedal, etc.) as part of their normal standard of care.

Exclusion Criteria:

* Subjects with a previous major amputation (at or above ankle)
* Subjects with end stage renal disease (ESRD) defined as significant renal dysfunction evidenced by estimated creatinine clearance of < 20 cc/min, or receiving chronic hemodialysis therapy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2001-08; Study Completion 2005-11

PRIMARY OUTCOMES:
Reduction in the proportion of subjects who experience a major amputation.
Reduction in proportion of subjects who die within 6 months from treatment initiation.

SECONDARY OUTCOMES:
Reduction in major amputation rate only.
Reduction in critical cardiovascular events (MI, stroke, CV death, etc.)
Improvement in graft patency of index operation.
Improvement in complete ulcer healing.
Improvement in pain at rest.
Improvement in quality of life.
Improvement in hemodynamic measurements.
Improvement in neuropathy.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (15):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Glendale, California
  - Los Angeles, California
  - San Francisco, California
  - Pensacola, Florida
  - Springfield, Illinois
  - Shawnee Mission, Kansas
  - Kenner, Louisiana
  - Royal Oak, Michigan
  - Biloxi, Mississippi
  - Rochester, New York
  - Durham, North Carolina
  - San Antonio, Texas
  - Tacoma, Washington
- United Kingdom (7):
  - Birmingham
  - Bristol
  - Dundee
  - Hull
  - London
  - Manchester
  - Southhampton